CLINICAL TRIAL: NCT04356898
Title: Glucose Profiles in Ramadan-fasting Diabetes Patients: Ramadan Flash Glucose Monitoring (RFGM) Study
Brief Title: Ramadan Flash Glucose Monitoring Study
Acronym: RFGM
Status: Completed | Type: Observational
Sponsor: Imperial College London Diabetes Centre (Other)
Responsible Party: Sponsor
Other Study IDs: IREC042
Record Dates: First submitted 2018-10-18; First posted 2020-04-22 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2018-10

CONDITIONS: Diabetes Mellitus
Keywords: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Diabetes fasting: Diabetes patients who decided to fast during the month of Ramadan
  Interventions: Other: No intervention
- Diabetes non-fasting: Diabetes patients who decided to not fast during the month of Ramadan
  Interventions: Other: No intervention
- Healthy: Healthy volunteers that decided to fast during the month of Ramadan
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Many Muslim patients with diabetes observe dawn to sunset fasting during the month of Ramadan. Hyperglycaemia and hypoglycaemia are possible problems amongst these patients. The aim of this study is to investigate glucose profiles in diabetes and non-diabetes patients that decided to fast or not to fast during Ramadan.

DETAILED DESCRIPTION:
A good knowledge of the profiles of blood glucose with different treatments can help in making Ramadan fasting free of unwanted effects for such patients. Previous studies, including the EPIDIAR have shown an increased risk of hypo- and hyperglycaemia in patients with diabetes who fast during the Holy month of Ramadan.Although self-monitoring of blood glucose (SMBG) is useful in fasting diabetes patients when used within a structured testing regimen, it requires a lot of effort and compliance from the patient and doesn't provide continuous blood glucose data. The amount of data provided using SMBG depends on the frequency of finger pricks measurements. Flash Glucose Monitoring (FGM) sensors provide a record of the individual's glucose levels, trends and patterns for up to 14 days. This sensor doesn't require calibration using finger pricks. FGM data show how day-to-day decisions and behaviours impact the control of blood sugar levels. Availability of FGM makes it possible to explore glucose profiles in a continuous fashion during Ramadan period and make comparisons with non-fasting times outside Ramadan. The aim of this study is to investigate glucose profiles in diabetes and non-diabetes patients that decided to fast or not to fast during Ramadan. The study will compare several parameters extracted from the FGM trace such us the incident of hypoglycaemia and hyperglycaemia, standard deviation, coefficient of variance and time in/above/below range. For this purpose the FreeStyle Libre sensor will be used. Patients will be asked to use the FreeStyle Libre sensor for a period of 3 months: 1 month before Ramadan, during Ramadan and one month after Ramadan.

ELIGIBILITY:
Inclusion Criteria:

* diabetes, age>=18

Exclusion Criteria:

* pregnancy, renal failure

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 321 (Actual)
Dates: Start 2018-04-15 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Change in mean glucose level; (mmol/L) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of change in mean glucose, in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).
Change in percentage of time in target blood glucose range (3.9 - 10.0 mmol/L); (%) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of change in percentage of time in target blood glucose range,in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).
Coefficient of variance (CV); (coefficient; no units) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of coefficient of variance of blood glucose, in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).
Area under the curve (AUC); ((mmol/L)*h) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of area under the curve for blood glucose, in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).

SECONDARY OUTCOMES:
Change in glucose management indicator (GMI) ; (index; no units) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of change in glucose management indicator (GMI) for blood glucose, in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).
Change in percentage of time in level 1 (<3.9 - 10.0 mmol/L) hypoglycaemic range (mmol/L); (%) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of change in percentage of time in level 1 hypoglycaemic range, in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).
Change in percentage of time in level 2 (<3.0 mmol/l) hypoglycaemic range (mmol/L); (%) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of change in percentage of time in level 1 hypoglycaemic range, in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).
Change in percentage of time in level 1 (>10.0 mmol/L); (%) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of change in percentage of time in level 1 hyperglycaemic range, in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).
Change in percentage of time in level 2 (>13.9 mmol/L); (%) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of change in percentage of time in level 1 hyperglycaemic range, in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).
Standard deviation (SD); (SD (no units) of glucose mmol/L) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of standard deviation of blood glucose, in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).
Low blood glucose index (LBGI) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of low blood glucose, in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).
High blood glucose index (HBGI) | Pre-Ramadan (30 days), Ramadan (29 days), Post-Ramadan (30 days)
  This primary outcome is aimed at measurement of high blood glucose, in patients with diabetes, at the time points/frames indicated (Pre-Ramadan, Ramadan and Post-Ramadan).

CONTACTS AND LOCATIONS:
Overall Officials: Nader Lessan, MD FRCP, Principal Investigator — Imperial College London Diabetes Center (ICLDC)
Locations (1):
- Imperial College London Diabetes Centre, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: No